CLINICAL TRIAL: NCT06821035
Title: Teaching Youth & Families Self-Regulation Skills to Disrupt the Impact of Adverse Childhood Experiences: Preventing Substance Use in Adversity- Impacted Youth
Brief Title: The THRIVE Study: Teaching Healthy Regulation in Individuals & Vulnerable Environments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other); University of Illinois at Chicago (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dawn Therese Bounds, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4821; 1R01DA060784-01 (NIH)
Record Dates: First submitted 2025-01-10; First posted 2025-02-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Adverse Childhood Experiences; Family Functioning
Keywords: Alcohol and Substance Use Prevention; Youth Risk Behaviors; Traumatized Youth; stress management; adolescent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GRIT Intervention (Experimental)
  Interventions: Behavioral: Garnering Resilience in Traumatized youth and families (GRIT)
- Digital Citizenship Curriculumn (Active Comparator)
  Interventions: Behavioral: Digital Citizenship Curriculum (DCC)

INTERVENTIONS:
Behavioral: Garnering Resilience in Traumatized youth and families (GRIT) — Dyads randomly assigned to Garnering Resilience in Traumatized youth and families (GRIT) will receive a community health worker delivered psychoeducational intervention that includes 6 weekly sessions focused on: 1) supportive health coaching to garner resilience via psychoeducation and the promotion of buffering protective factors in both youth and caregivers and 2) facilitating self-regulation using heart rate variability (HRV) biofeedback.
  Arms: GRIT Intervention
Behavioral: Digital Citizenship Curriculum (DCC) — Dyads randomly assigned to DCC will receive a community health worker-delivered, school grade-specific intervention that includes 6 weekly sessions focused on helping youth navigate the complexities of living in a digital world.
  Arms: Digital Citizenship Curriculumn

SUMMARY:
The goal of this 2-arm randomized control trial is to determine the impact of a community health worker delivered coaching intervention, GRIT, on preventing the early initiation of regular use of alcohol and cannabis among adversity-impacted adolescents ages 11-14 who do not regularly use alcohol or cannabis at baseline. The specific aims include:

* Aim 1. Examine the effect of GRIT on preventing the early initiation of regular alcohol and cannabis use over time.
* Aim 2. Examine the role of youth and caregiver self-regulation in mediating the effect of GRIT on adolescent rates of alcohol and cannabis use.

Researchers will compare participants who are randomized to the GRIT intervention to an active control group, receiving a Digital Citizenship Curriculum, to see if those who participate in GRIT experience greater improvements in self-regulation and lower cardiometabolic risks.

Participants will:

* Be randomized to either receive the GRIT intervention (experimental group) or the Digital Citizenship Curriculum (active control group)
* Complete 3 in-person visits at baseline, post-intervention, and 12-month post intervention
* Complete HRV assessments using emWave Pro Plus and survey assessments on REDCap during in-person visits.
* Participate in six 60-minute sessions conducted over 8 weeks via Zoom with an assigned community-health worker
* Be invited to complete a booster session at 6-months post-intervention
* Complete online measures at baseline, post-intervention, 6-month, and 12-month post-intervention

DETAILED DESCRIPTION:
Adverse Childhood Experiences (ACEs) constitute a serious public health issue, impacting almost half of adolescents and over 60% of adults in the United States. High ACEs exposure (i.e., four or more ACEs) may result in self-dysregulation (i.e., challenges managing cognitions, emotions, and behaviors) and lead to early initiation of alcohol and substance use (e.g., self-medication hypothesis) and other biopsychosocial responses, such as cardiometabolic risks (e.g., lowered heart rate variability [HRV], increased weight and blood pressure, and sleep disturbance), and emotional and/or cognitive dysregulation. Health inequities resulting from self-dysregulation are highest among minoritized and impoverished populations, who experience disproportionately higher exposure to ACEs, and early adolescence is a time in which experimentation with alcohol and drugs occurs. Although not all adolescents who experiment with drugs are later diagnosed with a substance use disorder, those who engage early (i.e., before the age of 14) and regularly are at greater risk. Youth with four or more ACEs may experience a unique type of adversity characterized by chronic, unpredictable stress shaping their perception of and responses to stress. However certain strategies, called Shift and Persist, can mitigate these exposures where one shifts their attention from adverse experiences to future-directed behaviors (e.g., healthy habit adoption, stress management), resulting in improved self-regulation and lower cardiometabolic risks. GRIT is a community health worker (CHW)-delivered psychoeducational health coaching intervention that promotes coping with high exposure to ACEs to regulate the stress response using self-regulation techniques and the development of healthy habits recommended by the California Surgeon General (e.g., supportive relationships, quality sleep, physical activity). We propose conducting a 2-arm Randomized Controlled Trial (RCT) (GRIT vs an active control [i.e., digital citizenship]) with 210 adolescent-caregiver dyads to determine GRIT's impact on preventing the early initiation of regular use of alcohol and cannabis among adversity-impacted adolescents ages 11-14 who do not regularly use alcohol or cannabis at baseline. The specific aims will: Aim 1. Examine the effect of GRIT on preventing the early initiation of regular alcohol and cannabis use over time. H1: Adolescents enrolled in GRIT will have lower rates of regular alcohol and/or cannabis use at post-intervention, 6-, and 12-month follow-ups compared to adolescents in the active control group. Aim 2. Examine the role of youth and caregiver self-regulation in mediating the effect of GRIT on adolescent rates of alcohol and cannabis use. H2: Youth and caregiver self-regulation will mediate youth initiation of regular alcohol and cannabis use. This community-based study seeks to establish efficacy for a brief, accessible secondary prevention program. Once efficacy is established and the mechanism of action is identified, larger confirmatory efficacy studies and effectiveness trials using innovative approaches (i.e. multi-family groups and social media) in additional settings offer the opportunity to scale and decrease the research-to-practice gap for adversity-impacted youth.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 11-14 years who score in the High-Risk category (i.e., 4 or more ACEs) on the ACEs and Toxic Stress Risk Assessment Algorithm
* Has access to a smartphone and is willing to download applicable apps (95% of all adolescents have access to a smartphone)
* Youth who are able to speak and read in English
* Has a parent/guardian/primary caregiver (18 years or older) who is English- or Spanish-speaking and willing to participate in the intervention.

Exclusion Criteria:

* Youth who cannot speak and read in English
* Youth who report any alcohol or cannabis use within the last 14 days
* Youth currently enrolled in another family-based intervention (i.e., family therapy)
* Youth in acute distress who are in immediate need of care (e.g., imminent risk of harm to self or others, active psychosis)
* Youth who report their caregivers' home environment is unsafe to return to, have been deemed unsafe, or require supervised visits by the Department of Children and Family Services (DCFS)
* Youth whose parent/guardian/primary caregiver declines participation will be referred to other programs in their community.
* Due to drug experimentation being common in adolescence, our interest in preventing the early initiation of regular use of alcohol and cannabis use, and youth who regularly use substances requiring a different intervention, we will enroll youth who initially report recent cannabis use but later report no use within the last two weeks and have a confirmatory negative urine drug screening.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol, Cannabis & Other Substance Use: CDC Youth Risk Behavior Surveillance System (YRBSS)+ Timeline Followback Method Assessment (TFB) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The YRBSS is a multiple-choice survey that collects health behavior history, including questions about alcohol and cannabis use. Youth who report any substance use in the last 30 days on the YRBS will complete the Timeline Followback Method Assessment (TFB) for the last 30 days. The TFB is used to assess recent marijuana, cigarette, alcohol and other drug use. The 14-item self-administered TFB asks respondents to retrospectively estimate their daily drug over a designated period of time, from 7 days to 2 years prior to the administration date. The TFB can be used to obtain a variety of quantitative estimates of substance use, including change in substance use. Predictive validity, concordance of the TFB with other measures of drug use and strong convergence among the TFB, urine assays, self-report and collateral parent and sibling reports have been demonstrated among white and minoritized adolescents.
Emotional Regulation: Difficulties in Emotional Regulation- Short Form (DERS-SF) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The DERS-SF is an 18-item abbreviated version of the original, 36-item DERS questionnaire. It measures emotion regulation ability based on 6 subscales: strategies, non-acceptance, impulse, goals, awareness, and clarity. All subscales on the DERS-SF are highly correlated with the original DERS, with correlations ranging from .91 -.98. Each of the DERS-SF subscales have a Cronbach α> .70 (ranging from .79 to .91). Total scores range from 18 to 90, with higher total score on the DERS-SF indicating greater difficulties in emotion regulation.

SECONDARY OUTCOMES:
Heart Rate Variability Assessment: EmWave Pro | Baseline, immediately after the intervention, 12 months post-intervention
  The emWave Pro is a heart rhythm monitoring system that helps to observe an individual's autonomic state. This software provides HRV assessments that can be used in a wide range of applications such as quantifying HRV levels. Using HeartMath's EmWAVE Pro software, every participant will have an HRV assessment conducted that includes a resting HRV assessment (3 minutes), a stress prep (3 minutes), and a 1-minute deep breathing assessment.
Sleep Quality: The Pittsburgh Sleep Quality Index (PSQI) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  PSQI is a 19-item questionnaire that assesses seven component scores; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The PSQI has an internal reliability of .83 and test-retest reliability of .85 for the global scale. PSQI global scores range from 0 to 21, with higher scores than 5 indicating sleep disturbance.
Nutrition: CDC Youth Risk Behavior Surveillance System (YRBSS) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The 2025 middle school version of the YRBSS is a national survey that includes 3 diet and weight-related items assessing nutrition that allow for national comparison with other youth.
Physical Activity: CDC Youth Risk Behavior Surveillance System (YRBSS) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The 2025 middle school version of the YRBSS is a national survey that includes 3 items assessing physical activity that allows national comparison with other youth.
Family Functioning: Family Assessment Device (FAD) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The FAD is a 60-item survey that assesses family functioning including problem solving, communication, roles, affective responsiveness, affective involvement, and behavior control. Scores range from 1 to 4 for each response. The higher the overall score, the worse the level of family function. It has reliability at .70 for all subscales except roles.
Psychological Flexibility: | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The Acceptance and Fusion Questionnaire (AFQ_Y8): an 8-item questionnaire developed for youth that examines their psychological inflexibility. It has an internal consistency of .83. Possible total scores range from 0 to 32. A higher total score indicates greater tendency to experience cognitive fusion (i.e. lower psychological flexibility).
Psychological Flexibility: | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The Acceptance and Action Questionnaire (AAQ-II): a 7-item questionnaire developed for adults to measure their psychological inflexibility and experimental avoidance. It has an internal consistency of .84 and test-retest reliability of .79- .81. Possible total scores range from 7 to 49. Higher total scores on the AAQ-II indicate higher psychological inflexibility, experiential avoidance, and more potential psychological distress. Lower total scores mean more psychological flexibility.
Psychological Stress: Perceived Stress Scale (PSS-10) | Baseline, immediately after the intervention, 6 months post-intervention, 12 months post-intervention
  The PSS-10 is a 10-item self-measure of psychological stress. It has two subscales: perceived helplessness & lack of self-efficacy. It has a Cronbach's alpha >.70 and a test-retest reliability of >.70. Total scores range from 0 to 40, with higher scores being indicative of higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn T. Bounds, Ph.D., Principal Investigator — University of California, Irvine; Norweeta G. Milburn, Ph.D., Study Director — University of California, Los Angeles; Karnik Niranjan, M.D., Ph.D., Study Director — University of California, Los Angeles; Shin Sanghyuk, Ph.D., Study Director — University of California, Irvine
Locations (1):
- The Regents of the University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be preserved using the National Addiction & HIV Data Archive Program (NAHDAP) repository within the Inter-university Consortium for Political and Social Research (ICPSR) platform. To protect participant privacy and confidentiality, shared data will be de-identified using participant ID's to designate each unique individual instead of names. Dates will be randomly shifted using REDCap. Data will be accompanied by detailed metadata to help ease of use. A DOI (Digital Object Identifier) will be assigned to our dataset, ensuring easy access and citation in future research.
Time Frame: At the time of publication or within 1 year of study completion.
Access Criteria: Data access will be restricted to individuals and institutions with clearly developed public health research objectives and mechanisms in place to oversee ethical use of the data. The restricted access process within NAHDAP will be used for this purpose.

REFERENCES:
- [Background] The prevalence of adverse childhood experiences, nationally, by state, and by race or ethnicity - Child Trends. ChildTrends. Accessed August 23, 2023.
- [Background] Nelson CA, Scott RD, Bhutta ZA, Harris NB, Danese A, Samara M. Adversity in childhood is linked to mental and physical health throughout life. BMJ. 2020 Oct 28;371:m3048. doi: 10.1136/bmj.m3048. PMID 33115717
- [Background] Giano Z, Wheeler DL, Hubach RD. The frequencies and disparities of adverse childhood experiences in the U.S. BMC Public Health. 2020 Sep 10;20(1):1327. doi: 10.1186/s12889-020-09411-z. PMID 32907569
- [Background] Anda RF, Felitti VJ, Bremner JD, Walker JD, Whitfield C, Perry BD, Dube SR, Giles WH. The enduring effects of abuse and related adverse experiences in childhood. A convergence of evidence from neurobiology and epidemiology. Eur Arch Psychiatry Clin Neurosci. 2006 Apr;256(3):174-86. doi: 10.1007/s00406-005-0624-4. Epub 2005 Nov 29. PMID 16311898
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Merrick MT, Ford DC, Ports KA, Guinn AS. Prevalence of Adverse Childhood Experiences From the 2011-2014 Behavioral Risk Factor Surveillance System in 23 States. JAMA Pediatr. 2018 Nov 1;172(11):1038-1044. doi: 10.1001/jamapediatrics.2018.2537. PMID 30242348
- [Background] Panisch LS, LaBrenz CA, Lawson J, et al. Relationships between adverse childhood experiences and protective factors among parents at-risk for child maltreatment. Child Youth Serv Rev. 2020;110:104816.
- [Background] Alabdulgader AA. Coherence: a novel nonpharmacological modality for lowering blood pressure in hypertensive patients. Glob Adv Health Med. 2012 May;1(2):56-64. doi: 10.7453/gahmj.2012.1.2.011. PMID 24278819
- [Background] Murray, Desiree W., Rosanbalm, Katie, Christopoulos, Christina, and Hamoudi, Amar. Self-Regulation and Toxic Stress: Foundations for Understanding SelfRegulation from an Applied Developmental Perspective. Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.; 2014.
- [Background] Khantzian EJ. The self-medication hypothesis of substance use disorders: a reconsideration and recent applications. Harv Rev Psychiatry. 1997 Jan-Feb;4(5):231-44. doi: 10.3109/10673229709030550. PMID 9385000
- [Background] Lloyd A, Brett D, Wesnes K. Coherence training in children with attention-deficit hyperactivity disorder: cognitive functions and behavioral changes. Altern Ther Health Med. 2010 Jul-Aug;16(4):34-42. PMID 20653294
- [Background] Suglia SF, Koenen KC, Boynton-Jarrett R, Chan PS, Clark CJ, Danese A, Faith MS, Goldstein BI, Hayman LL, Isasi CR, Pratt CA, Slopen N, Sumner JA, Turer A, Turer CB, Zachariah JP; American Heart Association Council on Epidemiology and Prevention; Council on Cardiovascular Disease in the Young; Council on Functional Genomics and Translational Biology; Council on Cardiovascular and Stroke Nursing; and Council on Quality of Care and Outcomes Research. Childhood and Adolescent Adversity and Cardiometabolic Outcomes: A Scientific Statement From the American Heart Association. Circulation. 2018 Jan 30;137(5):e15-e28. doi: 10.1161/CIR.0000000000000536. Epub 2017 Dec 18. PMID 29254928
- [Background] Hammond CJ, Chaney A, Hendrickson B, Sharma P. Cannabis use among U.S. adolescents in the era of marijuana legalization: a review of changing use patterns, comorbidity, and health correlates. Int Rev Psychiatry. 2020 May;32(3):221-234. doi: 10.1080/09540261.2020.1713056. Epub 2020 Feb 6. PMID 32026735
- [Background] Claypool N, Moore de Peralta A. The Influence of Adverse Childhood Experiences (ACEs), Including the COVID-19 Pandemic, and Toxic Stress on Development and Health Outcomes of Latinx Children in the USA: a Review of the Literature. Int J Child Maltreat. 2021;4(3):257-278. doi: 10.1007/s42448-021-00080-y. Epub 2021 Jul 11. PMID 34278229
- [Background] Maguire-Jack K, Lanier P, Lombardi B. Investigating racial differences in clusters of adverse childhood experiences. Am J Orthopsychiatry. 2020;90(1):106-114. doi: 10.1037/ort0000405. Epub 2019 Feb 28. PMID 30816722
- [Background] Chen E, McLean KC, Miller GE. Shift-and-Persist Strategies: Associations With Socioeconomic Status and the Regulation of Inflammation Among Adolescents and Their Parents. Psychosom Med. 2015 May;77(4):371-82. doi: 10.1097/psy.0000000000000157. PMID 26167560
- [Background] Volkow ND, Blanco C. Substance use disorders: a comprehensive update of classification, epidemiology, neurobiology, clinical aspects, treatment and prevention. World Psychiatry. 2023 Jun;22(2):203-229. doi: 10.1002/wps.21073. PMID 37159360
- [Background] Khurana A, Romer D, Betancourt LM, Brodsky NL, Giannetta JM, Hurt H. Experimentation versus progression in adolescent drug use: A test of an emerging neurobehavioral imbalance model. Dev Psychopathol. 2015 Aug;27(3):901-13. doi: 10.1017/S0954579414000765. Epub 2014 Aug 26. PMID 25154377
- [Background] Odgers CL, Caspi A, Nagin DS, Piquero AR, Slutske WS, Milne BJ, Dickson N, Poulton R, Moffitt TE. Is it important to prevent early exposure to drugs and alcohol among adolescents? Psychol Sci. 2008 Oct;19(10):1037-44. doi: 10.1111/j.1467-9280.2008.02196.x. PMID 19000215
- [Background] Flory K, Lynam D, Milich R, Leukefeld C, Clayton R. Early adolescent through young adult alcohol and marijuana use trajectories: early predictors, young adult outcomes, and predictive utility. Dev Psychopathol. 2004 Winter;16(1):193-213. doi: 10.1017/s0954579404044475. PMID 15115071
- [Background] Hingson RW, Heeren T, Winter MR. Age at drinking onset and alcohol dependence: age at onset, duration, and severity. Arch Pediatr Adolesc Med. 2006 Jul;160(7):739-46. doi: 10.1001/archpedi.160.7.739. PMID 16818840
- [Background] Sartor CE, Jackson KM, McCutcheon VV, Duncan AE, Grant JD, Werner KB, Bucholz KK. Progression from First Drink, First Intoxication, and Regular Drinking to Alcohol Use Disorder: A Comparison of African American and European American Youth. Alcohol Clin Exp Res. 2016 Jul;40(7):1515-23. doi: 10.1111/acer.13113. Epub 2016 Jun 3. PMID 27256613
- [Background] Murray DW, Rosanbalm K, Christopoulos C, Meyer AL. An Applied Contextual Model for Promoting Self-Regulation Enactment Across Development: Implications for Prevention, Public Health and Future Research. J Prim Prev. 2019 Aug;40(4):367-403. doi: 10.1007/s10935-019-00556-1. PMID 31372788
- [Background] Robson DA, Allen MS, Howard SJ. Self-regulation in childhood as a predictor of future outcomes: A meta-analytic review. Psychol Bull. 2020 Apr;146(4):324-354. doi: 10.1037/bul0000227. Epub 2020 Jan 6. PMID 31904248
- [Background] Nawi AM, Ismail R, Ibrahim F, Hassan MR, Manaf MRA, Amit N, Ibrahim N, Shafurdin NS. Risk and protective factors of drug abuse among adolescents: a systematic review. BMC Public Health. 2021 Nov 13;21(1):2088. doi: 10.1186/s12889-021-11906-2. PMID 34774013
- [Background] National Institute on Drug Abuse. NIDA Priority Scientific Area #2: Develop and Test Novel Prevention, Treatment, Harm Reduction, and Recovery Support Strategies. Published online 2022.
- [Background] Chen E, Miller GE. "Shift-and-Persist" Strategies: Why Low Socioeconomic Status Isn't Always Bad for Health. Perspect Psychol Sci. 2012 Mar;7(2):135-58. doi: 10.1177/1745691612436694. PMID 23144651
- [Background] Dormal V, Vermeulen N, Mejias S. Is heart rate variability biofeedback useful in children and adolescents? A systematic review. J Child Psychol Psychiatry. 2021 Dec;62(12):1379-1390. doi: 10.1111/jcpp.13463. Epub 2021 Jun 21. PMID 34155631
- [Background] Goessl VC, Curtiss JE, Hofmann SG. The effect of heart rate variability biofeedback training on stress and anxiety: a meta-analysis. Psychol Med. 2017 Nov;47(15):2578-2586. doi: 10.1017/S0033291717001003. Epub 2017 May 8. PMID 28478782
- [Background] Lehrer P, Kaur K, Sharma A, Shah K, Huseby R, Bhavsar J, Sgobba P, Zhang Y. Heart Rate Variability Biofeedback Improves Emotional and Physical Health and Performance: A Systematic Review and Meta Analysis. Appl Psychophysiol Biofeedback. 2020 Sep;45(3):109-129. doi: 10.1007/s10484-020-09466-z. PMID 32385728
- [Background] Goodrum NM, Prinz RJ. Family-Based Prevention of Child Traumatic Stress. Pediatr Clin North Am. 2022 Aug;69(4):633-644. doi: 10.1016/j.pcl.2022.04.011. PMID 35934490
- [Background] Hsiung H, Patel K, Hundal H, Baccouche BM, Tsao KW. Preventing Substance Abuse in Adolescents: A Review of High-Impact Strategies. Cureus. 2022 Jul 27;14(7):e27361. doi: 10.7759/cureus.27361. eCollection 2022 Jul. PMID 36046301
- [Background] Preventing Marijuana Use Among Youth | SAMHSA Publications and Digital Products. Accessed August 23, 2023.
- [Background] Chatterjee D, McMorris B, Gower AL, Forster M, Borowsky IW, Eisenberg ME. Adverse Childhood Experiences and Early Initiation of Marijuana and Alcohol Use: The Potential Moderating Effects of Internal Assets. Subst Use Misuse. 2018 Aug 24;53(10):1624-1632. doi: 10.1080/10826084.2017.1421224. Epub 2018 Jan 24. PMID 29364764
- [Background] Rioux C, Castellanos-Ryan N, Parent S, Vitaro F, Tremblay RE, Seguin JR. Age of Cannabis Use Onset and Adult Drug Abuse Symptoms: A Prospective Study of Common Risk Factors and Indirect Effects. Can J Psychiatry. 2018 Jul;63(7):457-464. doi: 10.1177/0706743718760289. Epub 2018 Apr 22. PMID 29682999
- [Background] Lander L, Howsare J, Byrne M. The impact of substance use disorders on families and children: from theory to practice. Soc Work Public Health. 2013;28(3-4):194-205. doi: 10.1080/19371918.2013.759005. PMID 23731414
- [Background] Gruber KJ, Taylor MF. A Family Perspective for Substance Abuse: Implications from the Literature. J Soc Work Pract Addict. 2006;6(1-2):1-29.
- [Background] Newton NC, Champion KE, Slade T, Chapman C, Stapinski L, Koning I, Tonks Z, Teesson M. A systematic review of combined student- and parent-based programs to prevent alcohol and other drug use among adolescents. Drug Alcohol Rev. 2017 May;36(3):337-351. doi: 10.1111/dar.12497. Epub 2017 Mar 23. PMID 28334456
- [Background] Kumpfer KL, Magalhães C. Strengthening Families Program: An Evidence-Based Family Intervention for Parents of High-Risk Children and Adolescents. J Child Adolesc Subst Abuse. 2018;27(3):174-179.
- [Background] Foxcroft DR, Ireland D, Lister-Sharp DJ, Lowe G, Breen R. Longer-term primary prevention for alcohol misuse in young people: a systematic review. Addiction. 2003 Apr;98(4):397-411. doi: 10.1046/j.1360-0443.2003.00355.x. PMID 12653810
- [Background] Burkhart K, Ievers-Landis CE, Huth-Bocks A. Introduction to the Special Issue on Adverse Childhood Experiences (ACEs): Prevention, Intervention, and Access to Care. Children (Basel). 2022 Aug 11;9(8):1205. doi: 10.3390/children9081205. PMID 36010095
- [Background] Christophe NK, Stein GL, Martin Romero MY, Chan M, Jensen M, Gonzalez LM, Kiang L. Coping and Culture: The Protective Effects of Shift-&-Persist and Ethnic-Racial Identity on Depressive Symptoms in Latinx Youth. J Youth Adolesc. 2019 Aug;48(8):1592-1604. doi: 10.1007/s10964-019-01037-8. Epub 2019 May 27. PMID 31134561
- [Background] McLaughlin KA, Lambert HK. Child Trauma Exposure and Psychopathology: Mechanisms of Risk and Resilience. Curr Opin Psychol. 2017 Apr;14:29-34. doi: 10.1016/j.copsyc.2016.10.004. PMID 27868085
- [Background] Hughes K, Bellis MA, Hardcastle KA, Sethi D, Butchart A, Mikton C, Jones L, Dunne MP. The effect of multiple adverse childhood experiences on health: a systematic review and meta-analysis. Lancet Public Health. 2017 Aug;2(8):e356-e366. doi: 10.1016/S2468-2667(17)30118-4. Epub 2017 Jul 31. PMID 29253477
- [Background] Chang X, Jiang X, Mkandarwire T, Shen M. Associations between adverse childhood experiences and health outcomes in adults aged 18-59 years. PLoS One. 2019 Feb 7;14(2):e0211850. doi: 10.1371/journal.pone.0211850. eCollection 2019. PMID 30730980
- [Background] Rothman EF, Edwards EM, Heeren T, Hingson RW. Adverse childhood experiences predict earlier age of drinking onset: results from a representative US sample of current or former drinkers. Pediatrics. 2008 Aug;122(2):e298-304. doi: 10.1542/peds.2007-3412. PMID 18676515
- [Background] Ford ES, Anda RF, Edwards VJ, Perry GS, Zhao G, Li C, Croft JB. Adverse childhood experiences and smoking status in five states. Prev Med. 2011 Sep;53(3):188-93. doi: 10.1016/j.ypmed.2011.06.015. Epub 2011 Jun 25. PMID 21726575
- [Background] Forster M, Gower AL, Borowsky IW, McMorris BJ. Associations between adverse childhood experiences, student-teacher relationships, and non-medical use of prescription medications among adolescents. Addict Behav. 2017 May;68:30-34. doi: 10.1016/j.addbeh.2017.01.004. Epub 2017 Jan 6. PMID 28088740
- [Background] Dube SR, Felitti VJ, Dong M, Chapman DP, Giles WH, Anda RF. Childhood abuse, neglect, and household dysfunction and the risk of illicit drug use: the adverse childhood experiences study. Pediatrics. 2003 Mar;111(3):564-72. doi: 10.1542/peds.111.3.564. PMID 12612237
- [Background] Brown MJ, Masho SW, Perera RA, Mezuk B, Cohen SA. Sex and sexual orientation disparities in adverse childhood experiences and early age at sexual debut in the United States: results from a nationally representative sample. Child Abuse Negl. 2015 Aug;46:89-102. doi: 10.1016/j.chiabu.2015.02.019. Epub 2015 Mar 21. PMID 25804435
- [Background] Choi NG, DiNitto DM, Marti CN, Choi BY. Association of adverse childhood experiences with lifetime mental and substance use disorders among men and women aged 50+ years. Int Psychogeriatr. 2017 Mar;29(3):359-372. doi: 10.1017/S1041610216001800. Epub 2016 Oct 26. PMID 27780491
- [Background] Afifi TO, Taillieu T, Salmon S, Davila IG, Stewart-Tufescu A, Fortier J, Struck S, Asmundson GJG, Sareen J, MacMillan HL. Adverse childhood experiences (ACEs), peer victimization, and substance use among adolescents. Child Abuse Negl. 2020 Aug;106:104504. doi: 10.1016/j.chiabu.2020.104504. Epub 2020 May 8. PMID 32402816
- [Background] Poudel A, Gautam S. Age of onset of substance use and psychosocial problems among individuals with substance use disorders. BMC Psychiatry. 2017 Jan 11;17(1):10. doi: 10.1186/s12888-016-1191-0. PMID 28077106
- [Background] Romm KF, Patterson B, Crawford ND, Posner H, West CD, Wedding D, Horn K, Berg CJ. Changes in young adult substance use during COVID-19 as a function of ACEs, depression, prior substance use and resilience. Subst Abus. 2022;43(1):212-221. doi: 10.1080/08897077.2021.1930629. Epub 2021 Jun 4. PMID 34086537
- [Background] Williams L, Clements-Nolle K, Lensch T, Yang W. Exposure to adverse childhood experiences and early initiation of electronic vapor product use among middle school students in Nevada. Addict Behav Rep. 2020 Feb 19;11:100266. doi: 10.1016/j.abrep.2020.100266. eCollection 2020 Jun. PMID 32467855
- [Background] Marques AH, Silverman MN, Sternberg EM. Evaluation of stress systems by applying noninvasive methodologies: measurements of neuroimmune biomarkers in the sweat, heart rate variability and salivary cortisol. Neuroimmunomodulation. 2010;17(3):205-8. doi: 10.1159/000258725. Epub 2010 Feb 4. PMID 20134204
- [Background] Quiñones M, Gold SN, Ellis A. Chapter 3 - Defining trauma, adversity, & toxic stress. In: Marsh AN, Cox LJ, eds. Not Just Bad Kids. Academic Press; 2022:67-101.
- [Background] Thayer JF, Lane RD. Claude Bernard and the heart-brain connection: further elaboration of a model of neurovisceral integration. Neurosci Biobehav Rev. 2009 Feb;33(2):81-8. doi: 10.1016/j.neubiorev.2008.08.004. Epub 2008 Aug 13. PMID 18771686
- [Background] Juster FT, Suzman R. An Overview of the Health and Retirement Study. J Hum Resour. 1995;30:S7-S56.
- [Background] Lee DY, Kim E, Choi MH. Technical and clinical aspects of cortisol as a biochemical marker of chronic stress. BMB Rep. 2015 Apr;48(4):209-16. doi: 10.5483/bmbrep.2015.48.4.275. PMID 25560699
- [Background] Adam EK, Quinn ME, Tavernier R, McQuillan MT, Dahlke KA, Gilbert KE. Diurnal cortisol slopes and mental and physical health outcomes: A systematic review and meta-analysis. Psychoneuroendocrinology. 2017 Sep;83:25-41. doi: 10.1016/j.psyneuen.2017.05.018. Epub 2017 May 24. PMID 28578301
- [Background] Thayer JF, Brosschot JF. Psychosomatics and psychopathology: looking up and down from the brain. Psychoneuroendocrinology. 2005 Nov;30(10):1050-8. doi: 10.1016/j.psyneuen.2005.04.014. PMID 16005156
- [Background] Schwerdtfeger AR, Schwarz G, Pfurtscheller K, Thayer JF, Jarczok MN, Pfurtscheller G. Heart rate variability (HRV): From brain death to resonance breathing at 6 breaths per minute. Clin Neurophysiol. 2020 Mar;131(3):676-693. doi: 10.1016/j.clinph.2019.11.013. Epub 2019 Dec 4. PMID 31978852
- [Background] Leyro TM, Buckman JF, Bates ME. Theoretical implications and clinical support for heart rate variability biofeedback for substance use disorders. Curr Opin Psychol. 2019 Dec;30:92-97. doi: 10.1016/j.copsyc.2019.03.008. Epub 2019 Apr 2. PMID 31055246
- [Background] Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Med Biol Eng Comput. 2006 Dec;44(12):1031-51. doi: 10.1007/s11517-006-0119-0. Epub 2006 Nov 17. PMID 17111118
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Visted E, Sorensen L, Osnes B, Svendsen JL, Binder PE, Schanche E. The Association between Self-Reported Difficulties in Emotion Regulation and Heart Rate Variability: The Salient Role of Not Accepting Negative Emotions. Front Psychol. 2017 Mar 9;8:328. doi: 10.3389/fpsyg.2017.00328. eCollection 2017. PMID 28337160
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] The Coherent Heart: Heart-Brain Interactions, Psychophysiological Coherence, and the Emergence of System-Wide Order. HeartMath Institute. Accessed August 23, 2023.
- [Background] Meyer PW, Muller LE, Zastrow A, Schmidinger I, Bohus M, Herpertz SC, Bertsch K. Heart rate variability in patients with post-traumatic stress disorder or borderline personality disorder: relationship to early life maltreatment. J Neural Transm (Vienna). 2016 Sep;123(9):1107-18. doi: 10.1007/s00702-016-1584-8. Epub 2016 Jun 16. PMID 27311838
- [Background] Schneider M, Schwerdtfeger A. Autonomic dysfunction in posttraumatic stress disorder indexed by heart rate variability: a meta-analysis. Psychol Med. 2020 Sep;50(12):1937-1948. doi: 10.1017/S003329172000207X. Epub 2020 Aug 28. PMID 32854795
- [Background] Trivedi GY, Saboo B, Singh RB, Maheshwari A, Sharma K, Verma N. Can Decreased Heart Rate Variability be a Marker of Autonomic Dysfunction, Metabolic Syndrome and Diabetes? J Diabetol. 2019;10(2):48.
- [Background] Jarczok MN, Koenig J, Wittling A, Fischer JE, Thayer JF. First Evaluation of an Index of Low Vagally-Mediated Heart Rate Variability as a Marker of Health Risks in Human Adults: Proof of Concept. J Clin Med. 2019 Nov 11;8(11):1940. doi: 10.3390/jcm8111940. PMID 31717972
- [Background] Minassian A, Geyer MA, Baker DG, Nievergelt CM, O'Connor DT, Risbrough VB; Marine Resiliency Study Team. Heart rate variability characteristics in a large group of active-duty marines and relationship to posttraumatic stress. Psychosom Med. 2014 May;76(4):292-301. doi: 10.1097/PSY.0000000000000056. PMID 24804881
- [Background] Simpkins CA, Simpkins AM. Neuroscience for Clinicians: Evidence, Models, and Practice. Springer Science & Business Media; 2012.
- [Background] Mather M, Thayer J. How heart rate variability affects emotion regulation brain networks. Curr Opin Behav Sci. 2018 Feb;19:98-104. doi: 10.1016/j.cobeha.2017.12.017. PMID 29333483
- [Background] Eddie D, Kim C, Lehrer P, Deneke E, Bates ME. A pilot study of brief heart rate variability biofeedback to reduce craving in young adult men receiving inpatient treatment for substance use disorders. Appl Psychophysiol Biofeedback. 2014 Dec;39(3-4):181-92. doi: 10.1007/s10484-014-9251-z. PMID 25179673
- [Background] Alayan N, Eller L, Bates ME, Carmody DP. Current Evidence on Heart Rate Variability Biofeedback as a Complementary Anticraving Intervention. J Altern Complement Med. 2018 Nov;24(11):1039-1050. doi: 10.1089/acm.2018.0019. Epub 2018 May 21. PMID 29782180
- [Background] Pizzoli SFM, Marzorati C, Gatti D, Monzani D, Mazzocco K, Pravettoni G. A meta-analysis on heart rate variability biofeedback and depressive symptoms. Sci Rep. 2021 Mar 23;11(1):6650. doi: 10.1038/s41598-021-86149-7. PMID 33758260
- [Background] Karavidas MK, Lehrer PM, Vaschillo E, Vaschillo B, Marin H, Buyske S, Malinovsky I, Radvanski D, Hassett A. Preliminary results of an open label study of heart rate variability biofeedback for the treatment of major depression. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):19-30. doi: 10.1007/s10484-006-9029-z. Epub 2007 Mar 1. PMID 17333315
- [Background] Siepmann M, Aykac V, Unterdorfer J, Petrowski K, Mueck-Weymann M. A pilot study on the effects of heart rate variability biofeedback in patients with depression and in healthy subjects. Appl Psychophysiol Biofeedback. 2008 Dec;33(4):195-201. doi: 10.1007/s10484-008-9064-z. Epub 2008 Sep 19. PMID 18807175
- [Background] Lin IM, Fan SY, Yen CF, Yeh YC, Tang TC, Huang MF, Liu TL, Wang PW, Lin HC, Tsai HY, Tsai YC. Heart Rate Variability Biofeedback Increased Autonomic Activation and Improved Symptoms of Depression and Insomnia among Patients with Major Depression Disorder. Clin Psychopharmacol Neurosci. 2019 May 31;17(2):222-232. doi: 10.9758/cpn.2019.17.2.222. PMID 30905122
- [Background] Beckham AJ, Greene TB, Meltzer-Brody S. A pilot study of heart rate variability biofeedback therapy in the treatment of perinatal depression on a specialized perinatal psychiatry inpatient unit. Arch Womens Ment Health. 2013 Feb;16(1):59-65. doi: 10.1007/s00737-012-0318-7. Epub 2012 Nov 25. PMID 23179141
- [Background] Tan G, Dao TK, Farmer L, Sutherland RJ, Gevirtz R. Heart rate variability (HRV) and posttraumatic stress disorder (PTSD): a pilot study. Appl Psychophysiol Biofeedback. 2011 Mar;36(1):27-35. doi: 10.1007/s10484-010-9141-y. PMID 20680439
- [Background] Ginsberg JP, Berry ME, Powell DA. Cardiac coherence and posttraumatic stress disorder in combat veterans. Altern Ther Health Med. 2010 Jul-Aug;16(4):52-60. PMID 20653296
- [Background] Zucker TL, Samuelson KW, Muench F, Greenberg MA, Gevirtz RN. The effects of respiratory sinus arrhythmia biofeedback on heart rate variability and posttraumatic stress disorder symptoms: a pilot study. Appl Psychophysiol Biofeedback. 2009 Jun;34(2):135-43. doi: 10.1007/s10484-009-9085-2. Epub 2009 Apr 25. PMID 19396540
- [Background] Reyes FJ. Implementing Heart Rate Variability Biofeedback Groups for Veterans with Posttraumatic Stress Disorder. Biofeedback. 2014;42(4):137-142.
- [Background] Schuman DL, Killian MO. Pilot Study of a Single Session Heart Rate Variability Biofeedback Intervention on Veterans' Posttraumatic Stress Symptoms. Appl Psychophysiol Biofeedback. 2019 Mar;44(1):9-20. doi: 10.1007/s10484-018-9415-3. PMID 30229543
- [Background] Science of the Heart. HeartMath Institute. Accessed August 23, 2023.
- [Background] May RW, Seibert GS, Sanchez-Gonzalez MA, Fincham FD. Self-regulatory biofeedback training: an intervention to reduce school burnout and improve cardiac functioning in college students. Stress. 2019 Jan;22(1):1-8. doi: 10.1080/10253890.2018.1501021. Epub 2018 Oct 20. PMID 30345850
- [Background] Lehrer P, Vaschillo B, Zucker T, et al. Protocol for Heart Rate Variability Biofeedback Training. Biofeedback. 2013;41(3):98-109.
- [Background] Thurstone C, Lajoie T. Heart rate variability biofeedback in adolescent substance abuse treatment. Glob Adv Health Med. 2013 Jan;2(1):22-3. doi: 10.7453/gahmj.2013.2.1.005. PMID 24381821
- [Background] Hassett AL, Radvanski DC, Vaschillo EG, Vaschillo B, Sigal LH, Karavidas MK, Buyske S, Lehrer PM. A pilot study of the efficacy of heart rate variability (HRV) biofeedback in patients with fibromyalgia. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):1-10. doi: 10.1007/s10484-006-9028-0. Epub 2007 Jan 12. PMID 17219062
- [Background] Pagaduan JC, Chen YS, Fell JW, Wu SSX. Can Heart Rate Variability Biofeedback Improve Athletic Performance? A Systematic Review. J Hum Kinet. 2020 Jul 21;73:103-114. doi: 10.2478/hukin-2020-0004. eCollection 2020 Jul. PMID 32774542
- [Background] McCraty R. Following the Rhythm of the Heart: HeartMath Institute's Path to HRV Biofeedback. Appl Psychophysiol Biofeedback. 2022 Dec;47(4):305-316. doi: 10.1007/s10484-022-09554-2. Epub 2022 Jun 22. PMID 35731454
- [Background] Elbers J, McCraty R. HeartMath approach to self-regulation and psychosocial well-being. J Psychol Afr. 2020;30(1):69-79.
- [Background] Murray DW, Rosanbalm K. Promoting Self-Regulation in Adolescents and Young Adults: A Practice Brief. OPRE Report 2015-82. Office of Planning, Research and Evaluation; 2017. Accessed September 4, 2023.
- [Background] Self-Regulation and Toxic Stress Report 3: A Comprehensive Review of Self-Regulation Interventions From Birth Through Young Adulthood | Frank Porter Graham Child Development Institute. Accessed August 23, 2023.
- [Background] Reff J, Baschnagel JS. The role of affective urgency and emotion regulation in vaping susceptibility. Addict Behav Rep. 2021 May 27;14:100355. doi: 10.1016/j.abrep.2021.100355. eCollection 2021 Dec. PMID 34136632
- [Background] Windle M, Haardorfer R, Getachew B, Shah J, Payne J, Pillai D, Berg CJ. A multivariate analysis of adverse childhood experiences and health behaviors and outcomes among college students. J Am Coll Health. 2018 May-Jun;66(4):246-251. doi: 10.1080/07448481.2018.1431892. Epub 2018 Mar 5. PMID 29405856
- [Background] Swedo EA, D'Angelo DV, Fasula AM, Clayton HB, Ports KA. Associations of Adverse Childhood Experiences With Pregnancy and Infant Health. Am J Prev Med. 2023 Apr;64(4):512-524. doi: 10.1016/j.amepre.2022.10.017. Epub 2023 Jan 23. PMID 36697281
- [Background] Academy on Violence and Abuse|AVA|ACE Study|Violence|Abuse|Education|Research|Resources. Accessed August 23, 2023.
- [Background] Javier JR, Hoffman LR, Shah SI; Pediatric Policy Council. Making the case for ACEs: adverse childhood experiences, obesity, and long-term health. Pediatr Res. 2019 Oct;86(4):420-422. doi: 10.1038/s41390-019-0509-2. Epub 2019 Jul 22. No abstract available. PMID 31330528
- [Background] Community Health Workers. Accessed August 23, 2023.
- [Background] Milburn NG, Iribarren FJ, Rice E, Lightfoot M, Solorio R, Rotheram-Borus MJ, Desmond K, Lee A, Alexander K, Maresca K, Eastmen K, Arnold EM, Duan N. A family intervention to reduce sexual risk behavior, substance use, and delinquency among newly homeless youth. J Adolesc Health. 2012 Apr;50(4):358-64. doi: 10.1016/j.jadohealth.2011.08.009. Epub 2011 Oct 26. PMID 22443839
- [Background] Bounds DT, Otwell CH, Melendez A, Karnik NS, Julion WA. Adapting a family intervention to reduce risk factors for sexual exploitation. Child Adolesc Psychiatry Ment Health. 2020 Feb 18;14:8. doi: 10.1186/s13034-020-00314-w. eCollection 2020. PMID 32099581
- [Background] Bounds DT, Winiarski DA, Otwell CH, Tobin V, Glover AC, Melendez A, Karnik NS. Considerations for working with youth with socially complex needs. J Child Adolesc Psychiatr Nurs. 2020 Nov;33(4):209-220. doi: 10.1111/jcap.12288. Epub 2020 Jul 20. PMID 32691491
- [Background] Bounds DT, Stiles-Shields C, Schueller SM, Odgers CL, Karnik NS. Ethical considerations for developing pediatric mhealth interventions for teens with socially complex needs. J Child Adolesc Psychiatr Nurs. 2023 Feb;36(1):7-16. doi: 10.1111/jcap.12396. Epub 2022 Sep 22. PMID 36134754
- [Background] Bounds DT, Rodrigues SM, Balsam D, Lennan N, Rodriguez KR, Milburn NG. Creating Space for Adolescents and Families With Lived Experience of Homelessness to Build Familial Empathy, Communication, and Emotional Regulation: A Qualitative Study of Facilitators of Implementation. J Psychosoc Nurs Ment Health Serv. 2024 Jan;62(1):27-35. doi: 10.3928/02793695-20230622-01. Epub 2023 Jul 3. PMID 37379121
- [Background] Bounds DT, Rodrigues SM, Milburn NG. Strengthening Families to Disrupt Intergenerational Health Inequities With Adolescents at Risk for Commercial Sexual Exploitation, Substance Use, and HIV. Am J Public Health. 2023 Jun;113(S2):S124-S128. doi: 10.2105/AJPH.2023.307284. No abstract available. PMID 37339412
- [Background] Babic A, Tokalic R, Cunha JAS, et al. Risk of bias in Cochrane systematic reviews: assessments of risk related to attrition bias are highly inconsistent. Published online July 11, 2018:366658.
- [Background] Childre DL, Martin H, Beech D. The HeartMath Solution: The Institute of HeartMath's Revolutionary Program for Engaging the Power of the Heart's Intelligence. Reprint edition. HarperOne; 2000.
- [Background] Bradley RT, McCraty R, Atkinson M, Tomasino D, Daugherty A, Arguelles L. Emotion self-regulation, psychophysiological coherence, and test anxiety: results from an experiment using electrophysiological measures. Appl Psychophysiol Biofeedback. 2010 Dec;35(4):261-83. doi: 10.1007/s10484-010-9134-x. PMID 20559707
- [Background] Full article: Ubuntu HeartMath programme efficacy for social coherence and work spirit: Preliminary evidence. Accessed August 23, 2023.
- [Background] Full article: Young, Black, successful, and homeless: examining the unique academic challenges of Black students who experienced homelessness. Accessed August 23, 2023.
- [Background] McCraty R, Atkinson M. Resilience Training Program Reduces Physiological and Psychological Stress in Police Officers. Glob Adv Health Med. 2012 Nov;1(5):44-66. doi: 10.7453/gahmj.2012.1.5.013. Epub 2012 Nov 1. PMID 27257532
- [Background] McCraty R, Zayas MA. Cardiac coherence, self-regulation, autonomic stability, and psychosocial well-being. Front Psychol. 2014 Sep 29;5:1090. doi: 10.3389/fpsyg.2014.01090. eCollection 2014. PMID 25324802
- [Background] Li WC, Zhang J, Kearney P, Braithwaite G. Psychophysical Coherence Training Regulating Air Traffic Controller's Heart Rate Variability and Resilience to Fatigue. In: Harris D, Li WC, eds. Engineering Psychology and Cognitive Ergonomics. Lecture Notes in Computer Science. Springer International Publishing; 2021:142-150.
- [Background] Bedell W, Kaszkin-Bettag M. Coherence and health care cost--RCA actuarial study: a cost-effectiveness cohort study. Altern Ther Health Med. 2010 Jul-Aug;16(4):26-31. PMID 20653293
- [Background] McCraty R, Atkinson M, Lipsenthal L, Arguelles L. New hope for correctional officers: an innovative program for reducing stress and health risks. Appl Psychophysiol Biofeedback. 2009 Dec;34(4):251-72. doi: 10.1007/s10484-009-9087-0. Epub 2009 May 23. PMID 19466540
- [Background] McCraty R, Barrios-Choplin B, Rozman D, Atkinson M, Watkins AD. The impact of a new emotional self-management program on stress, emotions, heart rate variability, DHEA and cortisol. Integr Physiol Behav Sci. 1998 Apr-Jun;33(2):151-70. doi: 10.1007/BF02688660. PMID 9737736
- [Background] McCraty R, Atkinson M, Tomasino D. Impact of a workplace stress reduction program on blood pressure and emotional health in hypertensive employees. J Altern Complement Med. 2003 Jun;9(3):355-69. doi: 10.1089/107555303765551589. PMID 12816624
- [Background] McCraty R, Atkinson M, Dispenza J. One-minute deep breathing assessment and its relationship to 24-h heart rate variability measurements. Heart Mind. 2018;2:70.
- [Background] Imm PS, Chinman M, Kulesza M, Hunter S, Acosta J. Evidence-Based Practices: Community-Based Interventions to Reduce Alcohol Use and Misuse. In: Leukefeld CG, Gullotta TP, eds. Adolescent Substance Abuse: Evidence-Based Approaches to Prevention and Treatment. Issues in Children's and Families' Lives. Springer International Publishing; 2018:333-377.
- [Background] California Surgeon General's Office. California Surgeon General's Playbook. Stress Relief for Caregivers and Kids during COVID-19.; 2019.
- [Background] Traub F, Boynton-Jarrett R. Modifiable Resilience Factors to Childhood Adversity for Clinical Pediatric Practice. Pediatrics. 2017 May;139(5):e20162569. doi: 10.1542/peds.2016-2569. PMID 28557726
- [Background] Uddin J, Alharbi N, Uddin H, Hossain MB, Hatipoglu SS, Long DL, Carson AP. Parenting stress and family resilience affect the association of adverse childhood experiences with children's mental health and attention-deficit/hyperactivity disorder. J Affect Disord. 2020 Jul 1;272:104-109. doi: 10.1016/j.jad.2020.03.132. Epub 2020 May 1. PMID 32379600
- [Background] Elam KK, Johnson SL, Ruof A, Eisenberg DTA, Rej PH, Sandler I, Wolchik S. Examining the influence of adversity, family contexts, and a family-based intervention on parent and child telomere length. Eur J Psychotraumatol. 2022 Jun 30;13(1):2088935. doi: 10.1080/20008198.2022.2088935. eCollection 2022. PMID 35789082
- [Background] Schaeffer K. Most U.S. teens who use cellphones do it to pass time, connect with others, learn new things. Pew Research Center. Accessed August 23, 2023.
- [Background] Costa E. New Report: ACEs BRFSS Data Report- An Overview of Adverse Childhood Experiences in California | California PACEs Action (CA) | PACEsConnection. California PACEs Action (CA). Published October 27, 2020. Accessed August 23, 2023.
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Wright A. REDCap: A Tool for the Electronic Capture of Research Data. J Electron Resour Med Libr. 2016;13(4):197-201.
- [Background] Thakur N, Hessler D, Koita K, Ye M, Benson M, Gilgoff R, Bucci M, Long D, Burke Harris N. Pediatrics adverse childhood experiences and related life events screener (PEARLS) and health in a safety-net practice. Child Abuse Negl. 2020 Oct;108:104685. doi: 10.1016/j.chiabu.2020.104685. Epub 2020 Sep 5. PMID 32898839
- [Background] R: A language and environment for statistical computing (ISBN 3-900051-07-0) - ScienceOpen. Accessed August 23, 2023.
- [Background] Cohen J, Mannarino AP. Disseminating and Implementing Trauma-focused CBT in community settings. Trauma Violence Abuse. 2008 Oct;9(4):214-26. doi: 10.1177/1524838008324336. PMID 18936280
- [Background] Cohen JA, Mannarino AP. Trauma-Focused Cognitive Behavioural Therapy for Children and Parents. Child Adolesc Ment Health. 2008 Nov;13(4):158-162. doi: 10.1111/j.1475-3588.2008.00502.x. Epub 2008 Aug 19. PMID 32847188
- [Background] Embracing Your Demons: an Overview of Acceptance and Commitment Therapy (Written by Russell Harris) - NYC Cognitive Behavioral, PLLC. Accessed August 23, 2023.
- [Background] Olsen JM, Nesbitt BJ. Health coaching to improve healthy lifestyle behaviors: an integrative review. Am J Health Promot. 2010 Sep-Oct;25(1):e1-e12. doi: 10.4278/ajhp.090313-LIT-101. PMID 20809820
- [Background] Digital Citizenship Curriculum | Common Sense Education. Accessed August 23, 2023.
- [Background] Singh HK, Kennedy GA, Stupans I. Competencies and training of health professionals engaged in health coaching: A systematic review. Chronic Illn. 2022 Mar;18(1):58-85. doi: 10.1177/1742395319899466. Epub 2020 Jan 16. PMID 31948276
- [Background] Oremus M, Sharafoddini A, Morgano GP, Jin X, Xie F. A Computer-Assisted Personal Interview App in Research Electronic Data Capture for Administering Time Trade-off Surveys (REDCap): Development and Pretest. JMIR Form Res. 2018 Jan 23;2(1):e3. doi: 10.2196/formative.8202. PMID 30684429
- [Background] Jarvelin-Pasanen S, Sinikallio S, Tarvainen MP. Heart rate variability and occupational stress-systematic review. Ind Health. 2018 Nov 21;56(6):500-511. doi: 10.2486/indhealth.2017-0190. Epub 2018 Jun 16. PMID 29910218
- [Background] Low A, McCraty R. Heart rate variability: New perspectives on assessment of stress and health risk at the workplace. Heart Mind. Published online 2018. Accessed August 23, 2023.
- [Background] Lai MHC. Bootstrap Confidence Intervals for Multilevel Standardized Effect Size. Multivariate Behav Res. 2021 Jul-Aug;56(4):558-578. doi: 10.1080/00273171.2020.1746902. Epub 2020 Apr 11. PMID 32279536
- [Background] Kreidler SM, Muller KE, Grunwald GK, Ringham BM, Coker-Dukowitz ZT, Sakhadeo UR, Baron AE, Glueck DH. GLIMMPSE: Online Power Computation for Linear Models with and without a Baseline Covariate. J Stat Softw. 2013 Sep;54(10):i10. doi: 10.18637/jss.v054.i10. PMID 24403868
- [Background] California Department Public Health, Injury and Violence Prevention Branch and the California Department of Social Services, Office of Child Abuse Prevention, California Essentials for Childhood Initiative, the University of California, Davis Violence Prevention Research Program, the University of California, Firearm Violence Research Center. Adverse Childhood Experiences Data Report: Behavioral Risk Factor Surveillance System (BRFSS), 20112017: An Overview of Adverse Childhood Experiences in California. ; 2020. California Department of Public Health and the California Department of Social Services; 2020.
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Zhao X, Lynch JG Jr, Chen Q. Reconsidering Baron and Kenny: Myths and Truths about Mediation Analysis. J Consum Res. 2010;37(2):197-206.
- [Background] O'Rourke HP, MacKinnon DP. Reasons for Testing Mediation in the Absence of an Intervention Effect: A Research Imperative in Prevention and Intervention Research. J Stud Alcohol Drugs. 2018 Mar;79(2):171-181. doi: 10.15288/jsad.2018.79.171. PMID 29553343
- [Background] Kamenetz A. Report: More Than Half Of U.S. Children Now Own A Smartphone By Age 11. NPR.
- [Background] Audrain-McGovern J, Lerman C, Wileyto EP, Rodriguez D, Shields PG. Interacting effects of genetic predisposition and depression on adolescent smoking progression. Am J Psychiatry. 2004 Jul;161(7):1224-30. doi: 10.1176/appi.ajp.161.7.1224. PMID 15229055
- [Background] Sobell LC, Sobell MB. Timeline Follow-Back. In: Litten RZ, Allen JP, eds. Measuring Alcohol Consumption: Psychosocial and Biochemical Methods. Humana Press; 1992:41-72.
- [Background] Bry BH, Krinsley KE. Booster sessions and long-term effects of behavioral family therapy on adolescent substance use and school performance. J Behav Ther Exp Psychiatry. 1992 Sep;23(3):183-9. doi: 10.1016/0005-7916(92)90035-h. PMID 1487536
- [Background] Waldron HB, Slesnick N, Brody JL, Turner CW, Peterson TR. Treatment outcomes for adolescent substance abuse at 4- and 7-month assessments. J Consult Clin Psychol. 2001 Oct;69(5):802-13. PMID 11680557
- [Background] Dillon FR, Turner CW, Robbins MS, Szapocznik J. Concordance among biological, interview, and self-report measures of drug use among African American and Hispanic adolescents referred for drug abuse treatment. Psychol Addict Behav. 2005 Dec;19(4):404-13. doi: 10.1037/0893-164X.19.4.404. PMID 16366812
- [Background] Mpofu JJ, Underwood JM, Thornton JE, Brener ND, Rico A, Kilmer G, Harris WA, Leon-Nguyen M, Chyen D, Lim C, Mbaka CK, Smith-Grant J, Whittle L, Jones SE, Krause KH, Li J, Shanklin SL, McKinnon I, Arrey L, Queen BE, Roberts AM. Overview and Methods for the Youth Risk Behavior Surveillance System - United States, 2021. MMWR Suppl. 2023 Apr 28;72(1):1-12. doi: 10.15585/mmwr.su7201a1. PMID 37104281
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Wortmann JH, Jordan AH, Weathers FW, Resick PA, Dondanville KA, Hall-Clark B, Foa EB, Young-McCaughan S, Yarvis JS, Hembree EA, Mintz J, Peterson AL, Litz BT. Psychometric analysis of the PTSD Checklist-5 (PCL-5) among treatment-seeking military service members. Psychol Assess. 2016 Nov;28(11):1392-1403. doi: 10.1037/pas0000260. Epub 2016 Jan 11. PMID 26751087
- [Background] Zapolski TCB, Rowe AT, Banks DE, Faidley M. Perceived Discrimination and Substance Use among Adolescents: Examining the Moderating Effect of Distress Tolerance and Negative Urgency. Subst Use Misuse. 2019;54(1):156-165. doi: 10.1080/10826084.2018.1512625. Epub 2018 Nov 5. PMID 30395759
- [Background] Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. J Psychopathol Behav Assess. 2004;26(1):41-54.
- [Background] Livheim F, Tengström A, Bond FW, Andersson G, Dahl J, Rosendahl I. Psychometric properties of the Avoidance and Fusion Questionnaire for Youth: A psychological measure of psychological inflexibility in youth. J Context Behav Sci. 2016;5(2):103-110.
- [Background] Swaim R, Stanley L. Psychometric Evaluation of the Parental Monitoring Short Scale (PMSS).; 2022.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Falk CF, Vogel TA, Hammami S, Miocevic M. Multilevel mediation analysis in R: A comparison of bootstrap and Bayesian approaches. Behav Res Methods. 2024 Feb;56(2):750-764. doi: 10.3758/s13428-023-02079-4. Epub 2023 Feb 22. PMID 36814007
- [Background] Hogan JW, Laird NM. Intention-to-treat analyses for incomplete repeated measures data. Biometrics. 1996 Sep;52(3):1002-17. PMID 8805765